CLINICAL TRIAL: NCT05788575
Title: Study of the Incidence of Surgical Site Infections (SSI) in a Large Teaching Hospital in Rome, Italy.
Brief Title: Study of the Incidence of Surgical Site Infections Developed by Patients Hospitalized in the Wards of a Large Teaching Hospital in Rome, Italy
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Laurenti Patrizia, Chief of the Complex Operative Unit of Hospital Hygiene, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 1956
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2023-03

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Procedure: surgery — any surgery that an inpatient has undergone

SUMMARY:
The surgical departments of the hospital were included in the study on a rotational basis over a period of 5 months. All patients undergoing surgery during this period were enrolled in the study.

The data collection in each department lasted 6 months (8 in the case of the use of prostheses) of which:

* 5 months of continuous survey of hospitalized patients
* 30 days of post-operative surveillance for all operations, 90 days for operations involving the use of prosthetic material Surveillance ends when a surgical site infection occurs, even if the event is prior to 30 or 90 days.

For each surgery, information was recorded such as the type of surgery, duration, ASA score, prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing surgery

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hospitalized patients undergoing surgery
Sampling Method: Probability Sample
Enrollment: 5424 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Incidence of surgical site infection | 30 days or 90 days (prosthesis)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario "A. Gemelli" IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No